CLINICAL TRIAL: NCT05378022
Title: Application of LiveSpo Navax in Treatment of Acute Respiratory Disease in Children Infected With Influenza Virus
Brief Title: Effects of Nasal-spraying LiveSpo Navax in Treatment of Influenza Virus in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Children's Hospital, Vietnam (Other)
Responsible Party: Principal Investigator, Tran Thanh Tu, Vice Director of International Center, Vietnam National Children's Hospital, National Children's Hospital, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020S-06.2; No. 441/BVNTW-VNCSKTE (Other: Vietnam National Children's Hospital)
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Acute Respiratory Tract Infections
Keywords: Influenza Virus (Flu); Acute Respiratory Tract Infections (ARTIs); Children; Nasal-spraying probiotics; Viral load; Co-infection bacteria; Cytokines; Bacillus spores
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Blind, randomized, and controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: LiveSpo Navax and placebo 0.9% NaCl physiological saline are indistinguishable regarding taste and smell. The color and turbidity of LiveSpo Navax suspension is unrecognizable to investigators except the PI and analyzer, nurses, patient's parents, and patients due to opaque plastic container.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Control group receives the routine treatment and uses 0.9% NaCl physiological saline:
  Routine treatment is as follows:
  * Oral administrative drugs: antipyretic paracetamol (Efferegant®); expectorant Carbocysteine (Carbothiol®); antiviral Oseltamivir phosphate (Tamiflu®); antibiotics e.g. cefotaxim (Goldcefo®), Amoxicillin / clavulanic acid (Augmentin®) based on the results of antibiotic susceptibility test.
  * Aerosol therapy: bronchodilator e.g. salbutamol (Ventolin ®️inhaler) or budesonide (Pulmicort ®️Respules).
  Interventions: Drug: 0.9% NaCl physiological saline
- Navax (Experimental): Navax group receives the routine treatment and uses NaCl 0.9% plus B. subtilis and B. clausii at 5 billion CFU/5 mL (LiveSpo®️ Navax):
  Routine treatment is as follows:
  Oral administrative drugs: antipyretic paracetamol (Efferegant®); expectorant Carbocysteine (Carbothiol®); antiviral Oseltamivir phosphate (Tamiflu®); antibiotics e.g. cefotaxime (Goldcefo®), Amoxicillin / clavulanic acid (Augmentin®) based on the results of antibiotic susceptibility test.
  - Aerosol therapy: bronchodilator e.g. salbutamol (Ventolin ®️inhaler) or budesonide (Pulmicort ®️Respules).
  Interventions: Combination Product: LiveSpo Navax

INTERVENTIONS:
Combination Product: LiveSpo Navax — In Vietnam, LiveSpo Navax is manufactured as a Class-A medical device product (Product declaration No.210001337/PCBA-HN) under manufacturing standards approved by Hanoi Health Department, Ministry of Health, Vietnam (Certificate No YT117-19) and ISO 13485:2016.
  Other Names: Registration number: No.210001337/PCBA-HN
  Arms: Navax
Drug: 0.9% NaCl physiological saline — Nasal-spraying 0.9% NaCl physiological saline is prepared by extracting 5 mL from 0.9% NaCl intravenous infusion 500 mL PP bottle (B.Braun, Germany, product declaration No. VD-32732-19), and then pouring it into the same opaque plastic spraying 10 mL-bottle that is used for LiveSpo Navax.
  Other Names: Registration number: VD-32723-19
  Arms: Control

SUMMARY:
Acute Respiratory Tract Infections (ARTIs) in children are common diseases, with influenza virus types A and B is one of the main causes of serious symptoms in young children. Although an influenza vaccine is available, influenza vaccination requires annual injections, which made it difficult for young children to get effectively immunized. Moreover, antiviral nucleotide drugs including Tamiflu (oseltamivir) are unsafe for young children and are recommended only for high-risk patients. Probiotics have emerged as promising safe candidates for supportive treatment of ARTIs and reduction of antibiotic dependence in recent years. Here, investigators propose that direct spraying of probiotics into the nose can be a fast and effective symptomatic treatment for ARTIs due to influenza virus.

The aim of the study about to evaluate the effectiveness of nasal-spraying probiotics containing spores of two bacterial strains, Bacillus subtilis and Bacillus clausii in preventing and supporting the treatment of children having acute respiratory symptoms due to influenza infection.

Study Population: sample size is 70. Description of Sites: the study is carried out at Vietnam National Children's Hospital.

Description of Study Intervention: totally 70 eligible patients are divided randomly into 2 groups (n = 35/group each): Patients in Control group received the routine treatment and three times per day 0.9% NaCl physiological saline while the patients in the Navax group received three times per day LiveSpo Navax in addition to the same standard of care treatment. The standard treatment regimen is 2-5 days but can be extended further depending on the severity of the patient's respiratory failure.

Study duration: 15 months

DETAILED DESCRIPTION:
Influenza virus types A and B is the common virus that causes Acute Respiratory Tract Infections (ARTIs) with a high risk of bronchiolitis for young children and infants. Influenza-infection symptoms range from mild fever, cough, runny nose, and wheezing to severe symptoms such as fast pulse, fast breathing, and respiratory failure. In a systematic review and meta-analysis of the global burden of seasonal influenza respiratory infections in young children, they estimated that 28.000 - 111.500 children under the age of 5 die as a result of influenza infections in 2008, of which 99% of these deaths occurred in developing countries. Influenza vaccination requires annual injections, which made it difficult for young children to get effectively immunized. Moreover, antiviral nucleotide drugs including Tamiflu (oseltamivir) are unsafe for young children and are recommended only for high-risk patients. Probiotics have emerged as promising safe candidates for supportive treatment of ARTIs and reduction of antibiotic dependence in recent years. However, the use of oral administrative probiotics as functional foods is effective only for mild symptoms and not applicable for Acute RTIs (ARTIs). Here, investigators propose that direct spraying of probiotics into the nose can be a fast and effective symptomatic treatment for ARTIs.

The objective was to investigate the symptomatic treatment effects of probiotic product LiveSpo Navax, as a liquid-suspension form containing Bacillus spores of safe B. subtilis ANA4 and B. clausii ANA39 strains, in children having acute respiratory diseases caused by influenza virus, investigators evaluation of improved efficacy and reduced treatment time of LiveSpo Navax in influenza-infected children; and measurement of changes in influenza viral load, co-infectious bacterial concentrations, and major cytokine indicators in the nasopharyngeal samples before and after 2 days using LiveSpo Navax.

Methods: A randomized, blind, and controlled clinical trial is conducted. The patient's parents are required to provide the following information about their children: full name, sex, age, obstetric history, vaccination history, and antibiotic use history… After informed consent, 70 patients with ARTIs due to influenza virus will be randomized into 2 groups (n = 35/group): the control group (named "Control" group) uses 0.9% NaCl physiological saline and an experimental group (named the "Navax" group) use the probiotics LiveSpo Navax. The patient is given a coded spray in the form of a blind sample to ensure the objectivity of the study. The clinical follow-up will be 5 days, nasopharyngeal samples will be collected at day 0 and day 2 to evaluate potential reductions in viral load and co-infection bacteria, as well as modulation of overreacted cytokine release and the presence of probiotic spores in the patient's nasal mucosa.

Real-time PCR for detection of microorganism in nasopharyngeal samples: semi-quantitative assays for measuring changes in influenza viral load and co-infection bacterial concentrations is conducted by the real-time RT-PCR/PCR routine protocol which has been standardized under ISO 15189:2012 criteria and used in Vietnam National Children's Hospital. Detection of B. subtilis ANA4 and B. clausii ANA39 are also conducted by real-time PCR SYBR Green that has been standardized under ISO 17025: 2017 standard and routinely in the Key Laboratory of Enzyme and Protein Technology, VNU University of Science.

ELISA assays for cytokine levels: pro-inflammatory cytokines levels (pg/mL) including interleukin (IL-6, IL-8) and TNF-alpha are quantified using an enzyme-linked immunosorbent assay kit (ELISA) according to the manufacturer's instructions.

During treatment, patients are monitored daily for typical clinical symptoms of Flu-induced respiratory tract infections, including runny nose, fever, dry rales, moist rales, body temperature (oC), oxymetry (SpO2) (%), pulse (beats/min), and breath (beats/min) until discharged. The patients' health conditions are observed by doctors and nurses, and their pieces of information are filled into medical records. During this study, parents' patients are asked to abstain from consumption for their children of other probiotics, either via nasal spray or oral administration, and refrain from cleaning nose for their children with other 0.9% NaCl physiological saline sprayers.

Data collection and statistical analysis: individual medical records are collected, and the patient's information is then gathered and systematized in a data set. The efficacy of LiveSpo Navax is evaluated and compared to 0.9% NaCl physiological saline based on the following clinical and sub-clinical criteria obtained in Navax and Control groups: (i) the symptomatic-relieving day; (ii) the reduction levels (2^△Ct) of influenza viral load and co-infection bacteria concentrations. △Ct for target genes is calculated as Ct (threshold cycle) at day 2 - Ct at day 0 while Ct of internal control is adjusted to be equal among all samples; (iii) the reduction levels of IL-6, IL-8, and TNF-alpha cytokines. The tabular analysis is performed on dichotomous variables using the χ2 test or Fisher's exact test when the expected value of any cell is below five. Continuous variables are compared using either the Wilcoxon test, t-test, or the Mann-Whitney test when data are not normally distributed. The correlations among the variables are assessed by Spearman's correlation analysis. Statistical and graphical analyses are performed on GraphPad Prism v8.4.3 software (GraphPad Software, CA, USA). The significance level of all analyzes is set at p < 0.05. P-values.

Expected outcomes: (i) LiveSpo Navax alleviates influenza-infection symptoms about 30% more effectively, as indicated by 90% of patients using LiveSpo Navax (Navax group) are symptom-free at day 2-5 of intervention depending on symptoms, compared to 60% of patients in Control group; (ii) Patients in Navax group has more significant reductions in influenza viral load (>10 fold) than patients in Control group at day 2 of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children (male/female) aged from 4 months to 7 years
* Admitted to hospital due to upper respiratory infection
* Influenza A and B positive by rapid test
* Parents of the pediatric patient agree to participate in the study, explain and sign the research consent form.

Exclusion Criteria:

* Newborn babies
* Having a history of drug allergies
* Need oxygen therapy
* Discharged before day 2
* Lost to follow-up
* Withdrawn from the trial
* Continuing in the trial but missing data
* Meeting the criteria for psychiatric disorders other than depression and/or anxiety.

Ages: 4 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with free respiratory symptoms | Day 0 to day 5
  Percentage (%) of influenza-infected patients with free respiratory symptoms including runny nose, fever, dry rales, moist rales, fast breath, and fast pulse

SECONDARY OUTCOMES:
Patient's breath | Day 0 to day 5
  Influenza-infected patient's breath (beats/min) before and after nasal-spraying
Patient's pulse | Day 0 and day 5
  Influenza-infected patient's pulse (beats/min) before and after nasal-spraying
Patient's temperature | Day 0 and day 5
  Influenza-infected patient's temperature (oC) before and after nasal-spraying
Patient's pulse oxygen (SpO2) | Day 0 to day 5
  Influenza-infected patient's pulse oxygen-SpO2 (%) before and after nasal-spraying
Influenza virus concentration | Day 0 and day 2
  Concentration of influenza virus in nasopharyngeal samples, as indicated by real-time RT-PCR threshold cycle (Ct) value
Co-infection bacterial concentrations | Day 0 and day 2
  Co-infection bacterial concentrations in nasopharyngeal samples, as indicated by real time PCR threshold cycle (Ct) values
Cytokines levels | Day 0 and day 2
  Levels (pg/mL) of tumor necrosis factor-α (TNF-α), interleukin-6 (IL-6), and interleukin-8 (IL-8) in nasopharyngeal samples

CONTACTS AND LOCATIONS:
Overall Officials: Tu T Tran, PhD. MD., Principal Investigator — International Center, Vietnam National Children's Hospital
Locations (1):
- International Center, Vietnam National Children's Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data or samples share that will be coded, with no PHI include. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a study protocol, informed consent form (ICF), clinical study peport (CSR). For more information or to submit a request, please contact clinicaltrial.probiotics@gmail.com

REFERENCES:
- [Background] Doyle JD, Campbell AP. Pediatric influenza and illness severity: what is known and what questions remain? Curr Opin Pediatr. 2019 Feb;31(1):119-126. doi: 10.1097/MOP.0000000000000721. PMID 30531402
- [Background] Sellers SA, Hagan RS, Hayden FG, Fischer WA 2nd. The hidden burden of influenza: A review of the extra-pulmonary complications of influenza infection. Influenza Other Respir Viruses. 2017 Sep;11(5):372-393. doi: 10.1111/irv.12470. PMID 28745014
- [Background] Dawood FS, Chaves SS, Perez A, Reingold A, Meek J, Farley MM, Ryan P, Lynfield R, Morin C, Baumbach J, Bennett NM, Zansky S, Thomas A, Lindegren ML, Schaffner W, Finelli L; Emerging Infections Program Network. Complications and associated bacterial coinfections among children hospitalized with seasonal or pandemic influenza, United States, 2003-2010. J Infect Dis. 2014 Mar 1;209(5):686-94. doi: 10.1093/infdis/jit473. Epub 2013 Aug 28. PMID 23986545
- [Background] Eccles R. Understanding the symptoms of the common cold and influenza. Lancet Infect Dis. 2005 Nov;5(11):718-25. doi: 10.1016/S1473-3099(05)70270-X. PMID 16253889
- [Background] COMMITTEE ON INFECTIOUS DISEASES. Recommendations for Prevention and Control of Influenza in Children, 2021-2022. Pediatrics. 2021 Oct;148(4):e2021053745. doi: 10.1542/peds.2021-053745. Epub 2021 Sep 7. PMID 34493538
- [Background] Bustinduy AL, Sutherland LJ, Chang-Cojulun A, Malhotra I, DuVall AS, Fairley JK, Mungai PL, Muchiri EM, Mutuku FM, Kitron U, King CH. Age-Stratified Profiles of Serum IL-6, IL-10, and TNF-alpha Cytokines Among Kenyan Children with Schistosoma haematobium, Plasmodium falciparum, and Other Chronic Parasitic Co-Infections. Am J Trop Med Hyg. 2015 May;92(5):945-51. doi: 10.4269/ajtmh.14-0444. Epub 2015 Mar 9. PMID 25758654
- [Background] Diaz PV, Valdivia G, Gaggero AA, Bono MR, Zepeda G, Rivas M, Uasapud P, Pinto RA, Boza ML, Guerrero J. Pro-Inflammatory Cytokines in Nasopharyngeal Aspirate From Hospitalized Children With Respiratory Syncytial Virus Infection With or Without Rhinovirus Bronchiolitis, and Use of the Cytokines as Predictors of Illness Severity. Medicine (Baltimore). 2015 Sep;94(39):e1512. doi: 10.1097/MD.0000000000001512. PMID 26426613
- [Background] Duvigneau S, Sharma-Chawla N, Boianelli A, Stegemann-Koniszewski S, Nguyen VK, Bruder D, Hernandez-Vargas EA. Hierarchical effects of pro-inflammatory cytokines on the post-influenza susceptibility to pneumococcal coinfection. Sci Rep. 2016 Nov 22;6:37045. doi: 10.1038/srep37045. PMID 27872472
- [Background] Vazquez Y, Gonzalez L, Noguera L, Gonzalez PA, Riedel CA, Bertrand P, Bueno SM. Cytokines in the Respiratory Airway as Biomarkers of Severity and Prognosis for Respiratory Syncytial Virus Infection: An Update. Front Immunol. 2019 Jun 4;10:1154. doi: 10.3389/fimmu.2019.01154. eCollection 2019. PMID 31214165
- [Background] Pandolfi E, Panera N, Alisi A, Carloni E, Russo L, Campagna I, Rizzo C, Concato C, Linardos G, Piccioni L, Jackson S, Villani A, Midulla F, Tozzi AE. Cytokine expression patterns in hospitalized children with Bordetella pertussis, Rhinovirus or co-infection. Sci Rep. 2021 May 26;11(1):10948. doi: 10.1038/s41598-021-89538-0. PMID 34040002
- [Background] Hu W, DeMarcus LS, Sjoberg PA, Robbins AS. Inactivated influenza vaccine effectiveness among department of defense beneficiaries aged 6 months-17 years, 2016-2017 through 2019-2020 influenza seasons. PLoS One. 2021 Aug 27;16(8):e0256165. doi: 10.1371/journal.pone.0256165. eCollection 2021. PMID 34450617
- [Background] Smith JR, Ariano RE, Toovey S. The use of antiviral agents for the management of severe influenza. Crit Care Med. 2010 Apr;38(4 Suppl):e43-51. doi: 10.1097/CCM.0b013e3181c85229. PMID 19935416
- [Background] Sugaya N, Tamura D, Yamazaki M, Ichikawa M, Kawakami C, Kawaoka Y, Mitamura K. Comparison of the clinical effectiveness of oseltamivir and zanamivir against influenza virus infection in children. Clin Infect Dis. 2008 Aug 1;47(3):339-45. doi: 10.1086/589748. PMID 18582202
- [Background] American Academy of Pediatrics Committee on Infectious Diseases. Antiviral therapy and prophylaxis for influenza in children. Pediatrics. 2007 Apr;119(4):852-60. doi: 10.1542/peds.2007-0224. PMID 17403862
- [Background] Nicholson KG, Aoki FY, Osterhaus AD, Trottier S, Carewicz O, Mercier CH, Rode A, Kinnersley N, Ward P. Efficacy and safety of oseltamivir in treatment of acute influenza: a randomised controlled trial. Neuraminidase Inhibitor Flu Treatment Investigator Group. Lancet. 2000 May 27;355(9218):1845-50. doi: 10.1016/s0140-6736(00)02288-1. PMID 10866439
- [Background] Oo C, Barrett J, Hill G, Mann J, Dorr A, Dutkowski R, Ward P. Pharmacokinetics and dosage recommendations for an oseltamivir oral suspension for the treatment of influenza in children. Paediatr Drugs. 2001;3(3):229-36. doi: 10.2165/00128072-200103030-00005. PMID 11310719
- [Background] Wooltorton E. Oseltamivir (Tamiflu) unsafe in infants under 1 year old. CMAJ. 2004 Feb 3;170(3):336. No abstract available. PMID 14757668
- [Background] Martin-Loeches I, van Someren Greve F, Schultz MJ. Bacterial pneumonia as an influenza complication. Curr Opin Infect Dis. 2017 Apr;30(2):201-207. doi: 10.1097/QCO.0000000000000347. PMID 27984245
- [Background] Slack MPE. The evidence for non-typeable Haemophilus influenzae as a causative agent of childhood pneumonia. Pneumonia (Nathan). 2017 Jun 25;9:9. doi: 10.1186/s41479-017-0033-2. eCollection 2017. PMID 28702311
- [Background] Dietl B, Henares D, Boix-Palop L, Munoz-Almagro C, Garau J, Calbo E. Related Factors to Streptococcus pneumoniae Invasive Infection and Clinical Manifestations: The Potential Role of Nasopharyngeal Microbiome. Front Med (Lausanne). 2021 Apr 20;8:650271. doi: 10.3389/fmed.2021.650271. eCollection 2021. PMID 33996857
- [Background] Harun AM, Noor NFM, Zaid A, Yusoff ME, Shaari R, Affandi NDN, Fadil F, Rahman MAA, Alam MK. The Antimicrobial Properties of Nanotitania Extract and Its Role in Inhibiting the Growth of Klebsiella pneumonia and Haemophilus influenza. Antibiotics (Basel). 2021 Aug 10;10(8):961. doi: 10.3390/antibiotics10080961. PMID 34439011
- [Background] Shahbazi R, Yasavoli-Sharahi H, Alsadi N, Ismail N, Matar C. Probiotics in Treatment of Viral Respiratory Infections and Neuroinflammatory Disorders. Molecules. 2020 Oct 22;25(21):4891. doi: 10.3390/molecules25214891. PMID 33105830
- [Background] Lehtoranta L, Pitkaranta A, Korpela R. Probiotics in respiratory virus infections. Eur J Clin Microbiol Infect Dis. 2014 Aug;33(8):1289-302. doi: 10.1007/s10096-014-2086-y. Epub 2014 Mar 18. PMID 24638909
- [Background] Rautava S, Salminen S, Isolauri E. Specific probiotics in reducing the risk of acute infections in infancy--a randomised, double-blind, placebo-controlled study. Br J Nutr. 2009 Jun;101(11):1722-6. doi: 10.1017/S0007114508116282. Epub 2008 Nov 6. PMID 18986600
- [Background] Anaya-Loyola MA, Enciso-Moreno JA, Lopez-Ramos JE, Garcia-Marin G, Orozco Alvarez MY, Vega-Garcia AM, Mosqueda J, Garcia-Gutierrez DG, Keller D, Perez-Ramirez IF. Bacillus coagulans GBI-30, 6068 decreases upper respiratory and gastrointestinal tract symptoms in healthy Mexican scholar-aged children by modulating immune-related proteins. Food Res Int. 2019 Nov;125:108567. doi: 10.1016/j.foodres.2019.108567. Epub 2019 Jul 21. PMID 31554075
- [Background] Kumpu M, Kekkonen RA, Kautiainen H, Jarvenpaa S, Kristo A, Huovinen P, Pitkaranta A, Korpela R, Hatakka K. Milk containing probiotic Lactobacillus rhamnosus GG and respiratory illness in children: a randomized, double-blind, placebo-controlled trial. Eur J Clin Nutr. 2012 Sep;66(9):1020-3. doi: 10.1038/ejcn.2012.62. Epub 2012 Jun 13. PMID 22692023
- [Background] Liu S, Hu P, Du X, Zhou T, Pei X. Lactobacillus rhamnosus GG supplementation for preventing respiratory infections in children: a meta-analysis of randomized, placebo-controlled trials. Indian Pediatr. 2013 Apr;50(4):377-81. doi: 10.1007/s13312-013-0123-z. PMID 23665598
- [Result] Wang X, Li Y, O'Brien KL, Madhi SA, Widdowson MA, Byass P, Omer SB, Abbas Q, Ali A, Amu A, Azziz-Baumgartner E, Bassat Q, Abdullah Brooks W, Chaves SS, Chung A, Cohen C, Echavarria M, Fasce RA, Gentile A, Gordon A, Groome M, Heikkinen T, Hirve S, Jara JH, Katz MA, Khuri-Bulos N, Krishnan A, de Leon O, Lucero MG, McCracken JP, Mira-Iglesias A, Moisi JC, Munywoki PK, Ourohire M, Polack FP, Rahi M, Rasmussen ZA, Rath BA, Saha SK, Simoes EA, Sotomayor V, Thamthitiwat S, Treurnicht FK, Wamukoya M, Yoshida LM, Zar HJ, Campbell H, Nair H; Respiratory Virus Global Epidemiology Network. Global burden of respiratory infections associated with seasonal influenza in children under 5 years in 2018: a systematic review and modelling study. Lancet Glob Health. 2020 Apr;8(4):e497-e510. doi: 10.1016/S2214-109X(19)30545-5. Epub 2020 Feb 20. PMID 32087815
- [Derived] Tran TT, Phung TTB, Tran DM, Bui HT, Nguyen PTT, Vu TT, Ngo NTP, Nguyen MT, Nguyen AH, Nguyen ATV. Efficient symptomatic treatment and viral load reduction for children with influenza virus infection by nasal-spraying Bacillus spore probiotics. Sci Rep. 2023 Sep 8;13(1):14789. doi: 10.1038/s41598-023-41763-5. PMID 37684332